CLINICAL TRIAL: NCT02558621
Title: Clinical Trial on Performance and Acceptance of a New Robotic Assistance System During Spinal Fusion Surgery
Brief Title: New Robotic Assistance System for Spinal Fusion Surgery
Acronym: AQrate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KB Medical SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AQrate01/2015
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Degenerative Disc Disease; Spinal Stenosis; Spondylolisthesis; Spondylosis
Keywords: Robotic Spinal Fusion Surgery
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis; Spondylolisthesis; Spondylosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device: AQrate Robotic Assistance System (Experimental): Precise positioning of surgical instruments and spinal implants during general spinal surgery.
  Interventions: Device: AQrate Robotic Assistance System

INTERVENTIONS:
Device: AQrate Robotic Assistance System — Robotic guidance during spinal fusion surgery

SUMMARY:
The main objectives of the study are to evaluate the acceptance into operating flow, performance and safety of the AQrate Robotic Assisted System during the spinal fusion surgery

DETAILED DESCRIPTION:
Based on the literature review of similar devices and on the pre-clinical tests performed with the AQrate System on bench and cadavers, the study is build around the following hypothesis:

1. The design and principle of operation of the AQrate System permits a correct integration in the surgical procedure flow thus enabling the surgeon to benefit from its advantages while not generating any additional operational difficulties
2. The stability and ease of use of the device will permit the surgeon to achieve any planned spinal fusion without requiring additional assistance from the medical staff compared to a conventional spinal fusion surgery.
3. A spinal fusion surgery procedure that is performed with the use of the AQrate System is similar to conventional spinal fusion surgery. If correctly used, no additional adverse event should be observed.
4. The exposure to x-ray should decrease as the need of intraoperative recheck of pedicle screws placed should be reduced
5. The precision of placement of pedicle screw should not be adversely affected by the use of the system compared to conventional spinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age from 18 years to 85 years) scheduled for spinal fusion surgery,
* Primary spinal surgery (It is the first surgery on this patient's spine)
* Patient is capable of complying with study requirements, and
* Patient is willing to provide a signed informed consent.

Exclusion Criteria:

* Pregnancy and lactation
* Simultaneous participation in other clinical studies
* Infection or malignancy
* Previous spondylodesis
* Previous spinal surgical procedures
* Neurologic diseases (e.g. Charcot-Marie Tooth, Guillain-Barre syndrome, cerebral palsy, neurofibroma)
* Spinal cord abnormalities with any neurologic symptoms or signs
* Paraplegia
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study.
* Patient cannot follow study protocol, for any reason
* Patient cannot or will not sign informed consent
* Patients in emergency situation, are not legally competent, cannot understand the situation,
* Pediatric patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
clinical acceptance of the performance of the AQrate Robotic Assistance System. | Day of surgery
  The acceptance of the performance of the AQrate System will be measured by scale given to total of 8 questions.

SECONDARY OUTCOMES:
Intraoperative exposure to radiation | Day of surgery
  Exposure of radiation in seconds from O-arm or other imaging system used during surgery
Accuracy of spinal screws placed | Within one month of surgery
  The assessment of the accuracy of pedicle screw will be evaluated post operatively on the CT scan, at discharge with the Gertzbein grading scale and copared to a freehand technique

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Denis Patet, MD, Principal Investigator — Clinic Genolier, Switzerland
Locations (2):
- Switzerland (2):
  - Clinic Genolier, Genolier, Canton of Vaud
  - Hôpital du Valais, Sion, Valais

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kostrzewski S, Duff JM, Baur C, Olszewski M. Robotic system for cervical spine surgery. Int J Med Robot. 2012 Jun;8(2):184-90. doi: 10.1002/rcs.446. Epub 2011 Dec 21. PMID 22190547